CLINICAL TRIAL: NCT01145716
Title: Exploration of Acute TFCC-injuries in Association With Distal Radius Fractures
Brief Title: Exploration of Wrist Soft Tissue Injuries Associated With Wrist Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Johan Scheer MD, County Council of Ostergotland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OC Linkoping TFCC volar expl; Dnr M200-08 Linkoping (Other: Linkoeping University/County Council Ostergotland)
Record Dates: First submitted 2010-05-04; First posted 2010-06-17 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2009-11

CONDITIONS: Triangular Fibrocartilage Complex Injuries
Keywords: TFCC injuries; Distal radius fractures
MeSH Terms: conditions — Wrist Fractures | interventions — Arthroscopy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgical exploration (Other): Descriptive
  Interventions: Procedure: Arthroscopy, surgery

INTERVENTIONS:
Procedure: Arthroscopy, surgery — Ulno-volar wrist approach to the TFCC

SUMMARY:
The purpose of this study is to describe and stage lesions of the triangular fibrocartilage complex (TFCC) in association with distal radius fractures. 20 patients with dorsally dislocated AO type A fractures of the distal radius with sufficient displacement (based of cadaveric data) will be included. After stability testing and wrist arthroscopy. The TFCC is explored through a volar incision and injuries were documented and repaired from this approach.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Distal radius fracture
* Displacement > 20 degrees of dorsal angulation

Exclusion Criteria:

* Previous significant wrist injury
* Declines to participate
* Ulnar styloid fracture at base or proximal to it

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Residual instability symptoms | Approx 2-6 months to include the patients that meet the inclusion criteria. They will be followed for 6 momths
  Mechanisms of injury are poorly previously described. This study will hopefully confirm cadeveric data. There is some evidence that patients might benefit from acute repair. Residual instability can be both ulnocarpal and radioulnar.

SECONDARY OUTCOMES:
Adverse events | Three months
  Patients that accept to participate will undergo exploration from a (new) ulnovolar approach. The study is purely descriptive. Patients are monitored for adverse events such as nerve injury and infection for 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lars E Adolfsson, Assoc prof, Principal Investigator — Linkopeing University, Sweden
Locations (1):
- Dept of orthopedics, Linköping, Sweden

REFERENCES:
- [Background] Lindau T, Hagberg L, Adlercreutz C, Jonsson K, Aspenberg P. Distal radioulnar instability is an independent worsening factor in distal radial fractures. Clin Orthop Relat Res. 2000 Jul;(376):229-35. doi: 10.1097/00003086-200007000-00031. PMID 10906880
- [Background] Lindau T, Arner M, Hagberg L. Intraarticular lesions in distal fractures of the radius in young adults. A descriptive arthroscopic study in 50 patients. J Hand Surg Br. 1997 Oct;22(5):638-43. doi: 10.1016/s0266-7681(97)80364-6. PMID 9752922
- [Background] Geissler WB, Fernandez DL, Lamey DM. Distal radioulnar joint injuries associated with fractures of the distal radius. Clin Orthop Relat Res. 1996 Jun;(327):135-46. doi: 10.1097/00003086-199606000-00018. PMID 8641057